CLINICAL TRIAL: NCT01157819
Title: Safety and Efficacy of Once-Daily Dosing of FoamOtic Cipro (0.3% Ciprofloxacin Otic Foam) Compared to Twice-Daily Dosing of Ciloxan (0.3% Ciprofloxacin Otic Solution) in Patients With Acute External Otitis
Brief Title: Safety and Efficacy of Once-Daily Dosing of FoamOtic Cipro Compared to Twice-Daily Dosing of Ciloxan Ear Drops in Patients With Acute External Otitis
Acronym: Once-a-day
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otic Pharma (Industry)
Responsible Party: Dr. Rodrigo Yelin (Study Director), Otic Pharma LTD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-002-000
Record Dates: First submitted 2010-07-04; First posted 2010-07-07 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-03

CONDITIONS: Otitis Externa; Otorhinolaryngologic Diseases; Ear Diseases; Otitis
Keywords: swimmer's ear; ear drops; ear foam; otic foam; ear infection; ear pain; ear inflammation
MeSH Terms: conditions — Otitis Externa; Otorhinolaryngologic Diseases; Ear Diseases; Otitis; Earache | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciloxan Ear Drops (Active Comparator): Ciloxan (Alcon, Inc.) Sterile Ophthalmic and Ear Drops
  Interventions: Drug: 0.3% Ciprofloxacin Ear Drops
- Foam Otic Cipro (Experimental): Patients randomized to this study arm will receive the experimental product
  Interventions: Drug: FoamOtic Cipro

INTERVENTIONS:
Drug: 0.3% Ciprofloxacin Ear Drops — 4 gtt b.i.d. for 7 days.
  Other Names: Ciloxan; Ciprofloxacin; Cipro
  Arms: Ciloxan Ear Drops
Drug: FoamOtic Cipro — 0.3% Ciprofloxacin Otic Foam, 1 application, q.d. for 7 days
  Other Names: Ciprofloxacin; Cipro
  Arms: Foam Otic Cipro

SUMMARY:
The purpose of this study is to assess the Safety and Efficacy of Foam Otic Cipro (0.3% Ciprofloxacin Otic Foam), used once-daily for 7 days for the treatment of Acute Diffuse Otitis Externa, compared to commercial ear drops used twice daily for 7 days.

DETAILED DESCRIPTION:
Acute otitis externa (AOE) is defined as a diffuse inflammation of the external ear canal, which may also involve the pinna and/or the tympanic membrane. AOE is one of the most common infections encountered by otolaryngologists, pediatricians and family physicians. Diagnosis of AOE requires rapid onset (generally within 48 hours) of symptoms and signs of ear canal inflammation which includes: A) otalgia (often severe), itching or fullness, sometimes accompanied by reduced hearing or jaw pain; B) tenderness of the tragus and/or pinna; and C) diffuse ear canal edema with or without erythema, sometimes accompanied by ear discharge.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older eligible to sign by themselves.
* Have a clinical diagnosis of Acute Otitis Externa based on clinical observation and of presumed bacterial origin.
* Intact tympanic membrane
* Unilateral Acute Otitis Externa

Exclusion Criteria:

* Known allergy or sensitivity to Ciprofloxacin or other quinolones.
* Clinical Diagnosis of chronic suppurative otitis media (CSOM), acute otitis media (AOM), involvement of middle ear effusion (MEE).
* Patient has the non intact tympanic membrane.
* Patient has a serious underlying disease.
* Patients with known history of immune dysfunction/deficiency and those receiving immunosuppressive therapy.
* Patients with history of Diabetes mellitus.
* Bilateral Acute Otitis Externa.
* Patients with more than 80% of the ear canal occluded.
* Pregnant or lactating patients.
* Overt fungal Acute Otitis Externa.
* Local ear canal abnormalities such as abscess, granulation or polyps.
* Congenital abnormalities of the external auditory canal or obstructive bony exostosis in the treated ear.
* Mastoid or other suppurative non-infectious ear disorder (e.g. cholesteatoma) in the treated ear.
* Seborrheic dermatitis or other dermatological conditions of the external auditory canal which would complicate evaluation.
* Current Infection requiring systemic antimicrobial therapy.
* Current or previous use of topical or oral antibiotics (within 3 days) or long-acting antibiotics (within 7 days).
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical cure confirmed by significant reduction or absence of the disease symptoms a) Otalgia, b) tenderness with movement of pinna, and c) edema/ear canal occlusion | within 7 days after completion of treatment that lasts 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yehudah Roth, MD, Principal Investigator — Edith Wolfson Medical Center
Locations (2):
- Israel (2):
  - Wolfson Medical Center, Holon
  - Bet Roter Clinic, Clalit Health Services, Holon